CLINICAL TRIAL: NCT05089305
Title: Effect of Inhalation Administration of Ozone Plasma on Lung Function and Inflammatory Parameters in Patients With Pulmonary Sequelae Associated With Coronavirus 19 Infection (SARS-COV-2)
Brief Title: Ozone Plasma on Lung Function and Inflammatory Parameters in Pulmonary Sequelae Associated With Coronavirus 19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Principal Investigator, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUCS-INTEC-OLFISA-001
Record Dates: First submitted 2021-10-14; First posted 2021-10-22 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Plasma ozone; COVID-19; SARS CoV 2; Lung function
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Open-ended, uncontrolled clinical trial in 35 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ozone plasma (Experimental): Patients will be provided with an ion-laden cold atmospheric plasma administration equipment from the company Fulgur Vitae Model 9000, they will also be given the necessary indications for the use of the equipment, which they must use for 5 minutes three consecutive times a day, every 6 hours, for two weeks. They will also be provided with an atmospheric oxygen meter, with the indication to keep the ppb below 0.07.
  Interventions: Drug: Ozone plasma

INTERVENTIONS:
Drug: Ozone plasma — Patients will be provided with an ion-laden cold atmospheric plasma administration equipment from the company Fulgur Vitae Model 9000, they will also be given the necessary indications, as well as recommendations on the use of the equipment, which they must use for 5 minutes three consecutive times a day, every 6 hours, for two weeks. They will also be provided with an atmospheric oxygen meter, with the indication to keep the ppb below 0.07. You must record in your diary the start time, end and eventualities (in case of presenting them).

SUMMARY:
The risk for the development of complications from COVID-19 occurs mainly in patients over 65 years of age, with obesity, arterial hypertension, chronic lung diseases and immunosuppression states. Since the persistence of radiological imaging correlates with physiological deterioration, these patients are likely to be at increased risk of parenchymal lung disease.

It is known that the administration of Ozone, in any of the three phases of COVID-19 infection, is useful in the management of acute disease, both for its viricidal and anti-inflammatory activity, however, in the convalescence stage when the persistence of sequelae that can severely affect the quality of life of patients is identified.

DETAILED DESCRIPTION:
The objective of this study is to evaluate whether the administration by inhalation of ozone plasma favorably modifies lung function and inflammatory parameters in patients with pulmonary sequelae associated with coronavirus 19 infection (SARS-COV-2). We will conduct an open-ended, uncontrolled clinical trial in 35 male and female patients, between 25-80 years of age with previous confirmed diagnosis of COVID-19 infection with negative nasopharyngeal polymerase chain reaction assay (PCR) test and without active disease, patients will also continue with their usual treatment. Clinical findings and laboratory and cabinet tests include a basal and 14-day metabolic and inflammatory profile, body weight, body mass index (BMI) and blood pressure will be determined during the initial and final visit, as well as respiratory parameters by pulmonary function tests (spirometry, TLCo) and performing the 6 min walk test in endless band with pre- and post-walk oximetry measurements at the beginning and end of the study. Adverse events to treatment will be documented. Statistical analysis: Mann-Whitney U test and Wilcoxon exact test. A p <0.05 shall be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 25-80 years
* Individuals without active disease with previous confirmed diagnosis of COVID-19 infection with negative nasopharyngeal PCR test
* With characteristic chest radiographic images compatible with lung infection, particularly interstitial pneumonitis with previous unburied glass patches, cobblestone or areas of consolidation (during active disease)
* Sign a letter of consent under information

Exclusion Criteria:

* Patients taking the following medicines: Ivermectin, azithromycin, corticosteroids, colchicine, chlorine dioxide, oral anticoagulants such as acenocoumarin, apixaban, rivaroxaban; bronchodilators such as β2-agonists such as salbutamol and derivatives, as well as inhaled anticholinergics of the ipratropium bromide type and derivatives.
* Patients who present medical difficulty or contraindication to perform the 6 km walk test in band
* Patients with a history of community-acquired pneumonia, pulmonary neoplasms, heart, renal, or hepatic failure

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-12-21 (Estimated)

PRIMARY OUTCOMES:
Lung Function | 14 days
  Respiratory parameters by pulmonary function tests (spirometry, TLCo) and performing the 6 min walk test in endless band with pre- and post-walk oximetry measurements at the beginning and end of the study.
Inflammatory parameters | 14 days
  Inflammatory parameters by C reactive protein (CPR), Tumoral Necrosis Factor alfa (TNFa) and Interleukin 6 (IL-6) measurements at the beginning and end of the study.

SECONDARY OUTCOMES:
Blood Biometrics | 14 days
  Blood Biometrics at the beginning and end of the study.
Oxygen saturation | 14 days
  Oxygen saturation at the beginning and end of the study.
Ferritin | 14 days
  Ferritin at the beginning and end of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Fernando Grover Paez, Guadalajara, Jalisco
  - Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No